CLINICAL TRIAL: NCT04157907
Title: Reflective Functioning and Psychotherapy Processes in Mentalization Based Therapy
Brief Title: Reflective Functioning and Psychotherapy Processes in MBT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Theresa Wilberg, senior consultant and professor, Oslo University Hospital
Other Study IDs: 2018/0519
Record Dates: First submitted 2019-11-01; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Mentalization-Based Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with borderline personality disorder: Patients with borderline personality disorder included in the MBT program
  Interventions: Behavioral: Mentalization based therapy

INTERVENTIONS:
Behavioral: Mentalization based therapy — Mentalization based therapy is a specialized treatment for patients with borderline personality disorder. The treatment program combines individual and group therapy, as well as psychoeducation

SUMMARY:
Borderline personality disorder (BPD) is a pervasive mental disorder characterized by emotional instability, self-destructive behavior, identity problems and unstable relationships. Persons with this disorder usually experience significant distress in terms of depression, anxieties, suicidal behavior, and difficulties in close relationships as well as with work- and social functioning. Recent research has found the prognosis of BPD to be better than previously assumed, and many patients improve from treatment.

Mentalization based therapy (MBT) is a specialized evidenced based therapy for patients with BPD. Like for other specialized treatments for this disorder, the outcome of therapy is typically variable, some patients respond well to treatment, whereas others respond less. It is therefore important to understand how treatment works in order to improve therapies and tailor treatment to individual patients.

Mentalizing is the ability to understand ourselves and others in terms of mental states, like intentions, feelings, desires, attitudes, and so on, or briefly; the ability to mind own and other's minds. Impaired mentalizing capacity is an assumed core aspect of BPD, underlying many of the symptoms of this disorder. MBT focuses on the patients mentalizing difficulties and is typically offered as a long-term combined treatment program comprising individual and group therapy, as well as psychoeducation. Several studies have documented positive effects of MBT in terms of reduced suicidal behavior, symptoms, interpersonal problems, medication, and health service use. It is assumed that such clinical improvement is made possible by helping the patients to develop their mentalizing abilities.

Yet, no study has investigated whether patients' mentalizing capacity changes during MBT, or to what degree outcome of MBT is mediated by improved mentalizing. Mentalizing is, however, a complex phenomenon and difficult to measure. Research in this area has been hampered by a lack of suitable methods. Mentalizing is usually operationalized as Reflective Functioning (RF) assessed by the RF Scale. The gold standard is to apply the RF Scale on the Adult Attachment Interview. However, this is a time consuming and costly method, and there is a need for testing other methods as well.

The overall aim of the project is to study treatment processes in MBT for patients with BPD. It focuses on patients' mentalizing difficulties before, during and at the end of therapy. Mentalizing is assessed using different methods. Our main research questions are:

1. To what degree does patients' level of RF change during MBT?
2. Is there a relationship between RF and outcome of MBT?
3. What is the relationship between RF and therapy processes in MBT?
4. Is it possible to identify in-session processes that promote mentalizing?
5. What is the clinical utility of various methods of RF assessment?

DETAILED DESCRIPTION:
BACKGROUND Borderline personality disorder (BPD) BPD is a pervasive mental disorder characterized by emotional instability, self-destructive behavior, identity problems and unstable interpersonal relationships. The disorder is associated with high levels of symptom distress, suicidal behavior, psychosocial impairment, and high rates of comorbid mental disorders such as mood, anxiety, and substance use disorders, as well as significant health service utilization and costs. Recent research has found the prognosis of BPD to be better than previously assumed. Yet, despite high rates of diagnostic remission many patients continue to have poor vocational and social functioning.

Several specialized and evidence based psychotherapies targeting characteristic BPD symptoms have been developed during the past decades, like Dialectical behavioral therapy, Transference focused therapy, Schema focused therapy and Mentalization based therapy. Across specific treatment approaches the outcome of therapy is typically variable, some patients respond well to treatment, whereas others respond less or even deteriorate. It is therefore important to understand how treatment works in order to improve therapies and tailor treatment to individual patients.

Mentalization based therapy (MBT) MBT is a manualized psychodynamic psychotherapy which focuses specifically on the patients' mentalizing difficulties. Mentalization is defined as the capacity to perceive human behavior as expressions of mental states, like thoughts, affects, dreams and intentions, and is usually operationalized as Reflective Functioning (RF) assessed by the RF Scale. Impaired mentalizing capacity is an assumed core aspect of BPD underlying characteristic features such as poor affect regulation, impulse control problems, and incoherent internal representations of self and others leading to unstable relationships and self- esteem. MBT is prototypically a combined treatment program comprising individual and group therapy, as well as psychoeducation. Several studies, including RCTs have documented positive effects of MBT in terms of reduced suicidal behavior, symptoms, interpersonal problems, medication, and health service use. There are also indications that MBT may be particularly helpful for more severely disturbed patients with extensive comorbidity.

Yet, no study has investigated whether patients' mentalizing capacity changes during MBT, or to what degree outcome of MBT is mediated by improved RF. One study found that outcome of two different treatment approaches (not MBT) differentially depended on patients' pretreatment levels of RF, indicating that RF may be a valuable variable for treatment selection and outcome. There are also indications that RF may improve during Transference focused therapy. However, there is a general lack of studies investigating the role of RF in the unfolding of psychotherapy processes and outcome of MBT. Thus, more studies are needed to gain knowledge of mechanisms of change in MBT.

RF and psychotherapy processes Common therapeutic factors are factors that are believed to function across different types of treatment, in contrast to specific factors which are seen as operating as part of specific therapies and interventions. An early good therapeutic alliance between patient and therapist is the most widely recognized common factor in individual therapies. The Working Alliance Inventory is an established method for assessment of therapeutic alliance in individual therapy. As to group therapies alliance to therapists and group members, as well as group cohesion are suggested as important common factors, but the evidence is not consistent. Assessment of therapeutic factors in groups is, however more complicated due to the many relationships in therapy groups. The Group Questionnaire is a promising empirically derived instrument intended to comprise important dimensions of a patient's relationship to his/her therapy group.

However, the relationship between common and specific therapeutic factors is debated, e.g., specific interventions and factors may be necessary for common factors to come into play. We don't know if specific factors in MBT stimulate alliance and outcome, or if there are other important processes operating. Research should investigate how patients' pretreatment or in-session RF influence the therapeutic alliance to the individual therapist or group, and to what degree interventions intended to stimulate mentalization have an influence on patients' experience of alliance. These are complex processes and other patient characteristic as well as therapeutic interventions must be taken into account when analyzing such processes.

Assessment of RF The gold standard for assessment of RF is the RF Scale applied on the Adult Attachment Interview (AAI) with patient's narratives of his/her experiences with early attachment figures. Yet, the specific mentalizing difficulties often seen in patients with BPD, is a temporary breakdown of mentalizing, particularly during emotional storms in current close relationships. One concern is therefore that RF based on the AAI may not be able to capture such mentalizing collapses. Concordantly, there is incipient evidence that RF based on the AAI may be rather trait like and slow to change. Researchers in this field are currently searching for additional methods for RF assessment. For instance, the RF Scale has been applied to transcripts of therapy sessions, capturing RF as a more fluctuating and state like phenomenon. So far this adaption has only been used on MBT sessions in a study of 15 patients with comorbid BPD and substance dependence.

To move forward in the understanding of RF and psychotherapy processes in more detail one should preferably apply different methods for RF assessment. A part of the present project is therefore to evaluate RF by three different methods based on 1) AAI , 2) in-session interactions, and 3) a specially developed interview focusing on episodes of temporary break down of mentalizing ability.

AIMS The overall aim of the project is to study psychotherapy processes in MBT for patients with BPD. It focuses on patients' mentalizing difficulties before, during and at the end of therapy. Mentalization is operationalized as RF and assessed using different methods. The projects aims to investigate the role of patients' RF for clinical outcome, change in RF during and across sessions, patient-therapist interactions promoting or hindering reflection, and other psychotherapy processes that might mediate treatment response. To render possible studies of more differentiated treatment responses the project includes a variety of outcomes, ranging from treatment attendance and dropout, clinical symptoms, personality related variables, global functioning, health service use, and rehabilitation support.

RESEARCH QUESTIONS

1. To what degree does patients' level of RF change during MBT?
2. Is there a relationship between RF and outcome of MBT?

   1. Does RF predict clinical outcome in MBT?
   2. Is outcome in MBT mediated by RF?
   3. Is change in RF associated with change in core BPD problems such as poor affect regulation, impulse control, and unstable relationships?
3. What is the relationship between RF and therapy processes in MBT?

   1. Is RF related to patients' experience of therapeutic alliance in individual and group therapy?
   2. Is RF related to early drop-out and treatment completion?
   3. How does patients' RF interact with other patient characteristics in influencing therapeutic alliance and outcome?
4. Is it possible to identify in-session processes that promote mentalizing?

   1. Does therapist adherence to MBT predict better patient in-session mentalizing or outcome?
   2. Which in-session processes, including therapist interventions, promote or impede patient mentalizing?
5. What is the clinical utility of various methods of RF assessment?

   1. What are the relationships between interview based RF scored on AAI, BPD domain specific RF scored on a specifically developed "Mentalization breakdown interview", and observer rated RF based on video recordings of individual therapy sessions?
   2. What is the relationship between the various RF assessment methods and intensity and frequency of mentalization breakdowns?
   3. Do the different RF assessment methods perform differently regarding prediction and mediation of clinical outcome?

The project will be conducted at the Personality Outpatient Unit, Section of Personality Psychiatry, Oslo University Hospital, which is specialized in the treatment of patients with personality disorders. Currently the unit focuses primarily on BPD. A maximum of sixty consecutively admitted patients with BPD or BPD traits, age 18-40 years, and 6-10 therapists from the ordinary staff will be included as participants after informed consent.

ELIGIBILITY:
Inclusion Criteria:

- Borderline personality disorder or significant borderline traits

Exclusion Criteria:

* patients with psychotic disorders as their main problem
* Asperger's syndrome/autism spectrum disorders
* low IQ
* unregulated bipolar I disorders as their main problem

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Patients with borderline personality disorder or significant borderline traits, who are treated in the MBT program at the Personality Outpatient Unit, Oslo University Hospital (OUH).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Work and Social Adjustments Scale, WSAS, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  Work and social adaption
Global Assessment of Functioning, GAF, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  psychosocial functioning
Patient Health Questionnaire, PHQ-9, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  depression
Patient Health Questionnaire, GAD-7, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  anxiety
Self-harm, self-report, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  Self-harm
Suicide attempts, self-report, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  Suicide attempts
Circumplex of Interpersonal Problems, CIP, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  interpersonal problems
Severity Index of Personality Problems, SIPP-118, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  personality functioning
Level of Personality Functioning Scale, LPFS BF, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  personality functioning
Difficulties in Emotion Regulation Scale, DERS, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  emotional regulation
Toronto Alexithymia Scale, TAS-20, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  alexithymia
Reflective functioning based on AAI, change from baseline to 3 months follow-up | 3 months follow-up
  reflective functioning
Reflective functioning based on the mentalization breakdown interview, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  reflective functioning
Reflective functioning based on therapy sessions, change during treatment | 6, 12, 18, 24, 30 and 36 months
  reflective functioning
Months in work or studies, self report, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  work functioning
Experiences in Close relationships, ECR, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  attachment
Suicide ideation, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  Suicide ideation

SECONDARY OUTCOMES:
Substance use (from AUDIT and DUDIT), change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  substance use
EuroQoL, EQ-5D, change during treatment and 3 months follow-up | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  quality of life
Modified Overt Aggression Scale (selected items), change during treatment and 3 months follow | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  aggression
Working Alliance Inventory, WAI, change during treatment | 6, 12, 18, 24, 30 and 36 months
  therapeutic alliance
Group Questionnaire, GQ, change during treatment | 6, 12, 18, 24, 30 and 36 months
  alliance in group therapy
Client Satisfaction Scale, CSS, change during treatment and 3 months follow | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  treatment satisfaction
Health service use / NAV contacts and support, change during treatment and 3 months follow | 6, 12, 18, 24, 30 and 36 months, and 3 months follow-up
  Health services, social support and benefits

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Wilberg, professor, Principal Investigator — Department of Research and Development, Oslo University Hospital
Locations (1):
- Personality Outpatient Unit, Section of Personality Psychiatry, Clinic for Mental Health and Addiction, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ulvestad DA, Johansen MS, Kvarstein EH, Pedersen G, Wilberg T. Minding mentalizing - convergent validity of the Mentalization Breakdown Interview. Front Psychiatry. 2024 Jun 21;15:1380532. doi: 10.3389/fpsyt.2024.1380532. eCollection 2024. PMID 38974920